CLINICAL TRIAL: NCT01402362
Title: Prevalence of Glucose Intolerance and Risk Factors in Ethiopian Immigrants in Israel; Follow-up Study.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Diabetes and Endocrinology Unit, Hillel Yaffe Medical Center
Other Study IDs: 56-2011
Record Dates: First submitted 2011-07-24; First posted 2011-07-26 (Estimated); Last update posted 2011-07-26 (Estimated); Status verified 2011-06

CONDITIONS: Diabetes Mellitus; Glucose Intolerance
Keywords: Ethiopians; Diabetes Mellitus; Glucose tolerance; Israel; Included in the year 2000 study
MeSH Terms: conditions — Diabetes Mellitus; Glucose Intolerance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Ethiopians participating in previous study, year 2000

SUMMARY:
High risk population: Screening for impaired glucose tolerance.

ELIGIBILITY:
Inclusion Criteria:

* Participation in the year 2000 study
* Signature of Informed Consent Form

Exclusion Criteria:

Pregnancy

-

Ages: 25 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Ethiopian immigrants to Israel living in Hadera.
Sampling Method: Non-Probability Sample
Enrollment: 550 (Estimated)
Dates: Start 2011-09

PRIMARY OUTCOMES:
Percent of patients with Diabetes Mellitus or impaired glucose tolerance | Day 1 of study

SECONDARY OUTCOMES:
Prevalence of hypertension and hyperlipidemia | Day 1 of study

CONTACTS AND LOCATIONS:
Locations (1):
- Diabetes and Endocrinology Unit, Hillel Yaffe MC, POB169, Hadera, Israel